CLINICAL TRIAL: NCT03953833
Title: Phase I Clinical Trial on the Safety, Tolerability, Pharmacokinetics of B003 in the Treatment of HER2-positive Recurrent or Metastatic Breast Cancer
Brief Title: B003 in Patients With HER2-positive Recurrent or Metastatic Breast Cancer
Acronym: B003-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B003-101
Record Dates: First submitted 2019-04-25; First posted 2019-05-17 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2022-10

CONDITIONS: HER2-positive Breast Cancer
Keywords: DLT; MTD; Safety; tolerability; HER2-positive; Recombinant Humanized Anti-HER2 Monoclonal Antibody

STUDY DESIGN:
Intervention Model Description: The study is divided into the dose escalation group and the dose expansion group. Dose escalation stage: treatment cycle is administered every 21days,the infusion is taken at the first day of each treatment cycle.Observation period of DLT is from day 1 to day 21 of the first treatment cycle.
  Dose expansion stage: treatment cycle is administered every 21days and could be administered continuously until the disease progresses or is intolerable.DLT is not accessed during this stage.
  Blind method: open Test range: Domestic test
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- recombinant anti-HER2 humanized monoclonal antibody conjugate (Experimental): Drug Name : Recombinant anti-HER2 humanized monoclonal antibody conjugate for injection R & D code: B003 Drug Type : Biological Products
  Interventions: Biological: Recombinant anti-HER2 humanized monoclonal antibody conjugate for injection.R&D code: B003.

INTERVENTIONS:
Biological: Recombinant anti-HER2 humanized monoclonal antibody conjugate for injection.R&D code: B003. — Usage: Intravenous infusion; Dose escalation stage: doses 0.6, 1.2, 2.4, 3.6, 4.8 mg / kg, 1-6subjects each. Dose expansion stage: 20 subjects are enrolled and take the recommended dose based on the result of dose escalation stage.
  Infusion time：90 minutes(90min-106min suggested) for the first time; if no infusion reaction happens, the follow-up time is adjusted to at least30 minutes(30min-40min suggested).Dose escalation stage: treatment cycle is administered every 21days,the infusion is taken at the first day of each treatment cycle.Observation period of DLT is the 21st day of the first treatment cycle.

SUMMARY:
To assess the safety and tolerability characteristics of B003 in HER2-positive patients with recurrent or metastatic breast cancer. The dose-limiting toxicity (DLT) is assessed and the maximum tolerated dose (MTD) is explored.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤ age ≤ 75 years old, female;
2. Histological or cytologically confirmed recurrent or metastatic breast cancer,Anti-HER2 treatment failure for recurrent or metastatic disease;
3. According to RECIST v 1.1, patients with measurable and/or unmeasurable lesions: 1) Patients with bone metastases, as long as the bone metastases have never received radiotherapy, and the primary tumours are available for HER2 detection and Biomarker analysis, which can be enrolled.
4. Female patients of childbearing age, patients and/or their partners should agree to use a highly effective non-hormonal contraceptive method or two effective non-hormonal contraceptive methods. Continue to use the appropriate contraceptive measures during the study period and at least 6 months after the last dose.

   * Electrocorticography (ECOG) physical state (PS) is 0-1 points;
   * Expected to survive for more than 3 months;
   * Understand and voluntarily sign the informed consent form.

Exclusion Criteria:

1. Previously received T-DM1 or same type of drug for treatment, previously used trastuzumab within 3 months before the trial, previously involved in other clinical trials within 4 weeks before the trial.
2. Known to be allergic to the study drug or its components;
3. Have received any anti-cancer trial medication within 28 days prior to the start of the trial;
4. Have received hormone treatment within 7 days before the trial.
5. Hematological toxicity caused by previous treatment CTCAE ≥ 2 persistence (except hemoglobin) (NCI-CTCAE version 4.03);
6. A third gap effusion with clinical symptoms that cannot be controlled by drainage or other methods.
7. The cumulative dose of anthracyclines used meets the following values: doxorubicin or liposomal doxorubicin >450 mg/m2; epirubicin >900 mg/m2; mitoxantrone >120 mg/m2; Idarubicin > 90 mg/m2. If another anthracycline or more than one anthracycline is used, the cumulative dose should not exceed the equivalent dose of doxorubicin 500mg/m2
8. Patients with other malignant tumors (cervical cancer of StageI B or lower that has been cured, non-invasive basal cells or squamous cell skin cancer, complete remission (CR) > 10 years of malignant melanoma, Except for other malignant tumors with complete remission (CR) > 5 years);
9. Laboratory abnormalities: 1) Neutrophil count <1.5×109/L, 2) Platelet count <100×109/L, 3) Hemoglobin <90 g/L, 4) Total bilirubin > 1.5 x upper limit of normal (ULN), 5) Alanine aminotransferase (ALT), aspartate aminotransferase (AST) > 2.5 × ULN, 6) Serum creatinine >1.5×ULN or creatinine clearance <50 mL/min;
10. Currently suffering from a serious and uncontrollable systemic disease (eg, clinically significant cardiovascular disease, lung disease, active infection, or metabolic disease);
11. Have a tendency to hemorrhage and thrombosis: 1) Any CTCAE 4.03 Level 2 bleeding event occurred within 2 months prior to screening, or CTCAE 4.03 Level 3 and above bleeding events within the first 6 months of screening; 2) A history of gastrointestinal bleeding within 6 months prior to screening or a clear tendency to gastrointestinal bleeding. Such as: esophageal varices with bleeding risk, local active ulcer lesions, fecal occult blood + +; 3) There is currently active bleeding or coagulopathy (PT>16s, activated partial thromboplastin time >43s, thrombin time)>21s, INR≥2.3, all of which need to be ruled out), have bleeding tendency or are receiving thrombolysis or anti- Coagulation therapy; 4) Patients need anticoagulant therapy with warfarin or heparin; 5) Patients need long-term antiplatelet therapy (eg aspirin, clopidogrel); 6) Thrombotic or embolic events in the past 6 months, such as: cerebrovascular accidents (including transient ischemic attacks), pulmonary embolism;
12. History of severe cardiovascular disease: 1) According to NYHA (New York Heart Association), current cardiac function classification: grade III or IV; 2) There is currently congestive heart failure and New York Heart Association cardiac function grade II and above; 3) A history of unstable angina or myocardial infarction within 6 months prior to screening; 4) There are currently arrhythmias requiring therapeutic intervention (patients taking beta-blockers or digoxin can be enrolled); 5) According to the current two-dimensional echocardiographic results, the left ventricular ejection fraction (LVEF) is <50%; 6) Have a history of LVEF falling below 40%, or have had symptomatic congestive heart failure when treated with anti-HER2; 7) There is currently poorly controlled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >100 mmHg); 8) Cardiac troponin I ≥ 0.2 ng/mL;
13. There is a history of moderate or severe dyspnea at rest due to advanced malignancies or their complications or severe pulmonary primary disease, or current continuous oxygen therapy is required;
14. Symptomatic brain metastases, depression or schizophrenia;
15. History of immunodeficiency, including: HIV-positive, or other acquired, congenital immunodeficiency disease, or a history of organ transplantation;
16. Hepatitis B (HBsAg and / or HBcAb positive, and peripheral blood hepatitis B virus DNA titer test results beyond the normal range of the research center), and / or hepatitis C patients;
17. Alcohol dependence, hormone dependence or drug abusers;
18. The investigator believes that there are other factors that are not suitable for the trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 30 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | through study completion, an average of 2 years
  The maximum tolerated dose (MTD) is operationally defined in toxicology as the highest daily dose of a chemical that does not cause overt toxicity in subjects
Dose-Limiting Toxicity | From day 1 to day 21 of treatment
  Some of the major toxic side effects are the main reasons limiting the continued increase in the dose of chemotherapy drugs, which are the dose-limiting toxicity of chemotherapy drugs.
Immunogenicity assessment | through study completion, an average of 2 years
  Sample positive rate and Individual positive rate of Anti-drug antibody(ADA)
Titer of ADA positive sample | through study completion, an average of 2 years
  a test to determine the level or degree of ADA positive samples and analyse the effect on the plasma concentration.
Pharmacokinetics measurement A | through study completion, an average of 2 year
  According to the detection of the serum concentration of B003 in plasma sample, the diagram of drug concentration-time for individual and each dose group could be concluded.
  Peak Plasma Time (Tmax)
Pharmacokinetics measurement B | through study completion, an average of 2 year
  According to the detection of the serum concentration of B003 in plasma sample, the diagram of drug concentration-time for individual and each dose group could be concluded.
  Peak Plasma Concentration (Cmax)
Pharmacokinetics measurement C | through study completion, an average of 2 year
  According to the detection of the serum concentration of B003 in plasma sample, the diagram of drug concentration-time for individual and each dose group could be concluded.
  half-life time
Pharmacokinetics measurement D | through study completion, an average of 2 year
  According to the detection of the serum concentration of B003 in plasma sample, the diagram of drug concentration-time for individual and each dose group could be concluded.
  Mean Residence Time( MRT)
Pharmacokinetics measurement E | through study completion, an average of 2 year
  According to the detection of the serum concentration of B003 in plasma sample, the diagram of drug concentration-time for individual and each dose group could be concluded.
  Area under the plasma concentration versus time curve (AUC)
Pharmacokinetics measurement F | through study completion, an average of 2 year
  According to the detection of the serum concentration of B003 in plasma sample, the diagram of drug concentration-time for individual and each dose group could be concluded.
  elimination rate constant
Pharmacokinetics measurement G | through study completion, an average of 2 year
  According to the detection of the serum concentration of B003 in plasma sample, the diagram of drug concentration-time for individual and each dose group could be concluded.
  clearance rate(CL/F)
Therapeutic Efficacy A | from date of start from the infusion of the first subject until the date after two treatments of the last subject, assessed up to 14 months.
  Objective Remission Rate (ORR): to be defined as the percentage of patients with complete response or partial response. Patients with CR or PR for the first evaluation will be confirmed after 4weeks. Patients without any evaluations are regarded as none-response.
Therapeutic Efficacy B | from date of start from the infusion of the first subject until the date after two treatments of the last subject, assessed up to 14 months.
  Disease Control rate(DCR): to be defined as the percentage of patients with complete response, partial response or stable disease.
Therapeutic Efficacy C | from the date when he patient has CR or PR to the first evaluation until the date when the patient has disease progression or death, assessed up to 14 months.
  Duration of response(DOR): to be defined as the duration from the first evaluation time when the patient has CR or PR to the first evaluation time when the patient has disease progression or death.
Therapeutic Efficacy D | from the date when he patient has CR or PR to the first evaluation until the date when the patient has disease progression or death, assessed up to 14 months.
  Progression-free survival:to be defined as the duration from the time of first infusion to the first recording time when the patient has disease progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Jiang, Principal Investigator — West China Hospital; Yongsheng Wang, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China